CLINICAL TRIAL: NCT05435079
Title: Research on a New Nursing Model of New High-flow Oxygen Inhalation Device to Improve Pulmonary Function in Patients With Respiratory Failure
Brief Title: Research on a NTHF to Improve Pulmonary Function in Patients With Respiratory Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: A2022088
Record Dates: First submitted 2022-05-14; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-04

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Before the start of the study, all enrolled patients were required to sign an informed consent form. Patients who met the inclusion criteria were divided into NTHF (observation group) and AIRVOTM2 (Fisher & Paykel, Auckland, New Zealand) group (control group) in a 1:1 ratio.
Who Masked: Outcomes Assessor
Masking Description: This study is a single-blind study. The researcher clearly defines the treatment group, but index evaluation, data collection and data statistics are completed by different trained researchers, and they don't know the specific grouping.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- new type of tracheotomy high-flow oxygen therapy (NTHF) (Experimental): NTHF (connect the oxygen suction tube, Venturi, Fisher & Paykel MR850 heated humidifier, RT308 breathing tube with humidification tank, airtight suction tube and tracheotomy in sequence from the output end of the automatic pressure-adjustable oxygen flow meter Catheter), adjust the MR850 to invasive automatic transmission, the temperature sensor automatically adjusts and maintains the gas temperature at the inlet of the tracheostomy catheter at 37°C according to the feedback temperature, and adjusts according to the gas outflow from the exhalation port of the patient's inspiratory phase. The gas flow rate of the oxygen therapy device is 40-60L/min. According to the monitored pulse oxygen saturation (SpO 2 ), the concentration of the venturi valve and the corresponding oxygen flow rate are adjusted to maintain the SpO 2 between 94% and 100%.
  Interventions: Device: high-flow oxygen therapy device for tracheotomized patients
- Respiratory Humidification Treatment（ AIRVO TM 2） (Active Comparator): AIRVOTM 2 (Fisher & Paykel, Auckland, New Zealand), connect the special breathing circuit, tracheostomy joint and tracheostomy tube in sequence from the output end of the oxygen flow meter. The gas outflow from the mouth is the standard, adjust the output gas flow rate of the therapy device to 40-60L/min, adjust the oxygen concentration according to the monitored pulse oxygen saturation (SpO 2 ), and maintain the SpO 2 between 94% and 100%. .
  Interventions: Device: high-flow oxygen therapy device for tracheotomized patients

INTERVENTIONS:
Device: high-flow oxygen therapy device for tracheotomized patients — From the output end of the automatic pressure-adjustable oxygen flow meter, connect the oxygen suction tube, Venturi, Fisher & Paykel MR850 heated humidifier, RT308 breathing tube with humidification tank, closed sputum suction tube and tracheostomy tube), Adjust the MR850 to invasive automatic transmission, the temperature sensor automatically adjusts and maintains the gas temperature at the inlet of the tracheostomy tube at 37°C according to the feedback temperature, and adjusts the oxygen therapy device according to the gas outflow from the exhalation port of the patient's inspiratory phase. The gas flow rate is 40-60L/min. According to the monitored pulse oxygen saturation (SpO 2 ), the concentration of the venturi valve and the corresponding oxygen flow rate are adjusted to maintain the SpO 2 between 94% and 100%.

SUMMARY:
Patients with respiratory failure have high morbidity and mortality. Long-term mechanical ventilation causes a high medical burden and cannot cure respiratory failure. Therefore, in-depth research on early weaning and oxygen therapy nursing mode is needed. Currently, studies on artificial airway high-flow oxygen therapy are limited. Studies have reported that oxygen inhalation devices that increase expiratory resistance produce flow-dependent positive airway pressure and lung volume effects that improve oxygenation and ventilation. It means that the innovation of oxygen therapy device may be a change The key to improving lung function and reducing mechanical ventilation in patients with respiratory failure.

The project team is committed to the innovation of high-flow oxygen therapy devices and the research on oxygen therapy care. In the early stage, the "New Artificial Airway High Flow Oxygen Therapy Device" was designed (NTHF), in 2018, the new technology and new projects were declared and approved to solve the problem of the flow rate of oxygen therapy devices. In the pre-test, 78 tracheotomy patients were observed using NTHF and respiratory humidification therapy device (AIRVOTM2 ) with high-flow oxygen therapy. As a result, NTHF was superior to AIRVOTM2 in improving airway humidification, oxygenation effect and cost, and published an article, which was approved in 2019 "Non-inferiority of humidification performance of a novel high-flow oxygen therapy device in oxygen therapy for tracheostomy-off-weaned patients. In 2021, it will be approved for the promotion of appropriate technologies for health and health in Guangdong Province. Relying on the high-level clinical key specialties of Guangdong Province, support with scientific research technology and financial support conditions.

Research hypothesis: NTHF has the physiological effects of increasing the positive expiratory pressure of artificial airway, alveolar ventilation, and humidification, and can improve the lung function of patients with respiratory failure after tracheotomy.

DETAILED DESCRIPTION:
1.1 Patients with respiratory failure have high morbidity and mortality. Long-term mechanical ventilation causes a high medical burden and cannot cure respiratory failure. Therefore, it is necessary to In-depth study of daily off-line and oxygen therapy nursing mode. Currently, studies on artificial airway high-flow oxygen therapy are limited. Studies have reported that increased expiratory resistance Oxygen inhalation devices produce flow-dependent positive airway pressure and lung volume effects that improve oxygenation and ventilation. It means that the innovation of oxygen therapy device may be a change.The key to improving lung function and reducing mechanical ventilation in patients with respiratory failure.

1.2 The project team is committed to the innovation of high-flow oxygen therapy devices and research on oxygen therapy care. In the early stage, the "New Artificial Airway High Flow Oxygen Therapy Device" was designed (NTHF), in 2018, the new technology and new projects were declared and approved to solve the flow rate problem of oxygen therapy devices ,observing 78 tracheotomized patients using NTHF and respiratory humidification therapy device (AIRVOTM2) Perform high-flow oxygen therapy. As a result, NTHF was superior to AIRVOTM2 in improving airway humidification, oxygenation, and cost, and published an article. Approved in 2019 "New high-flow oxygen therapy device in tracheotomy Non-inferiority study of humidification performance in oxygen therapy for weaned patients" (funded 150,000 yuan, China Clinical Research Registry, ChiCTR1900023421). 2021 , it was approved to promote the "Artificial Airway High Flow Oxygen Therapy Airtight Suction Technology" in Guangdong Province for Health and Health Appropriate Technology . Relying on Guangdong Province High-level clinical key specialties,support with scientific research technology and financial support condition.

1.3 Scientific assumption: NTHF has the physiological effects of increasing positive expiratory pressure of artificial airway, alveolar ventilation, and humidification, and can improve respiratory failure trachea,The patient's lung function was incised.

2 goals 2.1 To evaluate the effect of NTHF on improving pulmonary ventilation, ventilation and defense function in patients with respiratory failure artificial airway.

2.2 Obtain evidence that NTHF improves pulmonary function in patients with respiratory failure, and establish a new model of oxygen therapy nursing for patients with artificial airway in respiratory failure.

3 Research content 3.1 In a randomized parallel control method, NTHF and AIRVOTM2 were used in two groups of patients with respiratory failure artificial airway, and the two groups of patients were observed for 7 days.

The oxygenation index, respiratory rate, and mechanical ventilation time were analyzed, and the improvement of oxygenation in patients with respiratory failure by two oxygen therapy devices was analyzed.

3.2 Comparing the results of pulmonary function tests and microbial metagenomic testing of the two groups of patients before treatment and after 7 days of treatment, to explore the effect of NTHF on improving pulmonary function and patient comfort in patients with mild and moderate respiratory failure, and to explore the effect of NTHF in patients with respiratory failure caused by different diseases. A new model of oxygen therapy care.

4 Key issues to be addressed 4.1 To verify the effect of the new high-flow oxygen therapy device in improving oxygenation, ventilation and humidification of patients with respiratory failure artificial airway.

4.2 To explore whether the new high-flow oxygen therapy device can improve the lung function of patients with respiratory failure artificial airway, and establish a new model of oxygen therapy nursing.

5 Expected results 5.1 Academic indicators: Establish a personalized weaning scheme for patients with respiratory failure and a new nursing model for tracheotomy and high-flow humidified oxygen therapy. Published papers 1-2Participate in academic exchange conferences.

5.2 Talent training: train 1-2 respiratory therapists and graduate students. 5.3 Social and economic benefits: reduce the time of mechanical ventilation in patients with respiratory failure,Shorten the days of hospitalization, reduce costs, and reduce the burden on families and society.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who ≥18 years old and meets the diagnostic criteria for respiratory failure
2. Have an artificial airway, ready or have been released from the ventilator
3. The circulation is basically stable, and there are no shocks of various types that are difficult to correct (mean arterial pressure remains unchanged under the condition of vasoactive drugs).

   <65mmHg)
4. Consciousness and ability to cooperate with clinical treatment

Exclusion Criteria:

1. Pregnancy and end-stage cancer patients
2. History of airway injury, pulmonary trauma, and lung surgery
3. Central respiratory failure or status asthmaticus caused by neurological diseases
4. Refusing to cooperate with treatment or to participate in the researcher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Level of oxygenation | 24hours after start of high flow oxygen therapy
  Oxygenation is assessed by arterial blood gas sample
Level of oxygenation | 48 hours after start of high flow oxygen therapy
  Oxygenation is assessed by arterial blood gas sample
Level of oxygenation | 7th days after start of high flow oxygen therapy
  Oxygenation is assessed by arterial blood gas sample

SECONDARY OUTCOMES:
level of sputum viscosity | 24th, 48th and 7th days after start of high flow oxygen therapy
  sputum viscosity is assessed with a sputum viscometer
Patient satisfaction scoreg greater than or equal to 90 | the 7th day after start of high flow oxygen therapy
  Using Hospital Designated Satisfaction Questionnaire which include comfort, bloating, dry mouth, ability to hear and speak（Total score is 100 points）

CONTACTS AND LOCATIONS:
Overall Officials: MEI YANGMEI, Study Chair — Shenzhen Second People's Hospital
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No